CLINICAL TRIAL: NCT04070027
Title: Progressive Resistance Training Versus Total Hip Arthroplasty in Patients With End-stage Hip Osteoarthritis (PROHIP): A Multicentre, Parallel-group, Randomised Controlled Superiority Trial
Brief Title: Progressive Resistance Training Versus Total Hip Arthroplasty in Patients With Hip Osteoarthritis
Acronym: PROHIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Odense University Hospital (Other); Naestved Hospital (Other); Aarhus University Hospital (Other); The Danish Rheumatism Association (Other); Region of Southern Denmark (Other); Association of Danish Physiotherapists (Other); The Research Council at Naestved-Slagelse-Ringsted Hospitals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-20180158; R153-A4771 (Other Grant/Funding Number: The Danish Rheumatism Association); R161-A5280 (Other Grant/Funding Number: The Danish Rheumatism Association); R166-A5553 (Other Grant/Funding Number: The Danish Rheumatism Association); R176-A6231 (Other Grant/Funding Number: The Danish Rheumatism Association); 18/41994 (Other Grant/Funding Number: The Region of Southern Denmark); 17/33622 (Other Grant/Funding Number: The Region of Southern Denmark)
Record Dates: First submitted 2019-08-12; First posted 2019-08-28 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Hip Osteoarthritis
Keywords: Total Hip Arthroplasty; Total Hip Replacement; Exercise; Progressive Resistance Training; Strength Training; Hip Joint
MeSH Terms: conditions — Osteoarthritis, Hip; Motor Activity | interventions — Arthroplasty, Replacement, Hip; Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Hip Arthroplasty (Active Comparator): A standard fast-track multimodal surgical program comprising patient information, optimised pain management, and early mobilisation. Total hip arthroplasty (THA) will be performed by experienced orthopaedic surgeons in accordance with the standard posterior surgical approach. Patients will receive standard postoperative rehabilitation consisting of either a standard leaflet with a hospital-specific home-based exercise program aimed at increasing hip muscle strength and range of motion or, if considered necessary, a referral to supervised hip-specific exercise therapy delivered at private physiotherapist clinics or municipal rehabilitation. Furthermore, postsurgical procedures will follow hospital-specific procedures ranging from no postsurgical control to postsurgical assessment of the hip and rehabilitation at the physiotherapy department (after six-weeks).
  Interventions: Procedure: Total Hip Arthroplasty
- Progressive Resistance Training (Active Comparator): A 12-week supervised explosive-type progressive resistance training (PRT) program with two training sessions a week. All training sessions will be conducted in municipal rehabilitation centres with one-to-one supervision and ≥48 hours of rest in between sessions. The standardised PRT program will consist of warm-up on a stationary bicycle (10 min) followed by four lower extremity exercises (50 min). Exercises will be performed unilaterally with as full range of motion as possible in sets of three separated by 60 sec of rest in the following order: leg press, hip extension, hip flexion, and hip abduction. Patients will be instructed to complete the concentric phase of each repetition "as fast as possible", maintain full extension for 1 sec, and perform the eccentric phase in 2-3 sec. Hip-related pain up to 5 rated on a Numerical Rating Scale (0-10) is considered acceptable during exercises. After the 12-weeks, patients will be offered three-months of optional unsupervised PRT.
  Interventions: Other: Progressive Resistance Training

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — Total hip arthroplasty following standard procedures.
  Other Names: Total Hip Replacement
  Arms: Total Hip Arthroplasty
Other: Progressive Resistance Training — Progressive resistance training based on available evidence on patients with hip osteoarthritis and designed in accordance with the "American College of Sports Medicine" (ACSM) recommendations for progression models in resistance training aiming at inducing muscle hypertrophy and increasing muscle strength and power.
  Other Names: Strength Training; Exercise
  Arms: Progressive Resistance Training

SUMMARY:
Hip osteoarthritis is associated with joint pain, physical disability, decreased muscle strength and poor health status, and the most common cause for total hip arthroplasty. No studies have investigated the effect of total hip arthroplasty compared to non-surgical treatment in patients with end-stage hip osteoarthritis. This comparison is of upmost importance as it is unknown whether non-surgical treatment may be used as an alternate to surgery.

The purpose of this study is to investigate whether total hip arthroplasty followed by standard care is superior to progressive resistance training for improving hip function and pain in patients with end-stage hip osteoarthritis.

The hypothesis is that patients treated with total hip arthroplasty will improve more than patients treated with progressive resistance training.

DETAILED DESCRIPTION:
Hip osteoarthritis (OA) is associated with joint pain, dysfunction of activities of daily living (ADL), decreased muscle strength and decline in health-related quality of life status, and the most common cause for total hip arthroplasty (THA). In Denmark, approximately 10.400 primary THA surgeries are performed annually, and the yearly incidence rate of this procedure has increased dramatically from 80 to 180 per 100.000 persons between 1995 and 2016. However, some patients experience long-term pain and may never recover full physical function and muscle strength after surgery.

Exercise has been shown to improve physical function and reduce pain in people with hip OA, and is recommended initially as a treatment in international clinical guidelines. Furthermore, a recent randomised controlled trial (RCT) showed clinically relevant improvements in ADL and muscle function after 10-weeks of supervised explosive-type progressive resistance training (PRT) in patients with end-stage hip OA scheduled for THA compared to standard preoperative care.

To date, no RCTs have investigated the effect of THA followed by standard postoperative care compared to supervised explosive-type PRT in patients with end-stage hip OA. Therefore, this highlights the need for a high-quality trial as it is unknown whether non-surgical treatment may be used as an alternate to surgery.

The aim of this randomised controlled trial is to investigate whether THA followed by standard care is superior to a 12-week supervised explosive-type PRT programme for improving patient-reported hip function and pain 6 months after initiating the intervention, measured using the Oxford Hip Score (OHS), in patients with end-stage hip OA eligible for THA. Exploratory outcome time-points will be assessed at 3, 12, 24 and 60 months after initiating the intervention.

The hypothesis is that THA followed by standard care is superior to a 12-week supervised explosive-type PRT programme for improving patient-reported hip function and pain 6 months after initiating the intervention, measured using the OHS, in patients with end-stage hip OA eligible for THA.

Observational cohort:

Patients fulfilling the eligibility criteria but declining to participate in the RCT will be asked to participate in a prospective observational cohort study using the same primary end-point (6 months), exploratory time-points (3, 12, 24 and 60 months), and patient-reported outcomes, but following usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥50 years
2. Clinical history and symptoms consistent with primary hip osteoarthritis (including hip osteoarthritis due to mild hip dysplasia that may be treated with standard components) and radiographic verified hip osteoarthritis defined as joint space narrowing <2 mm
3. Considered eligible for total hip arthroplasty by an orthopaedic surgeon (i.e. duration of symptoms >3 months, hip related pain, functional impairment or decreased range of motion (ROM), and attempted treatment with analgesics)

Exclusion Criteria:

1. Severe walking deficits (dependency of two crutches or walker)
2. Body Mass Index >35 kg/m2
3. Lower extremity fractures within one-year prior to inclusion
4. Planned other lower extremity surgery within six months
5. Cancer diagnosis and receiving chemo-, immuno- or radiotherapy
6. Neurological diseases (e.g. previous stroke, multiple sclerosis, Parkinson's, Alzheimer's).
7. Other reasons for exclusion (i.e. inadequacy in written and spoken Danish, mentally unable to participate, physically unable to comply with the PRT protocol due to comorbidity (e.g. severe heart disease, previous major lower extremity surgery within six-months) etc.).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in the Oxford Hip Score (OHS) from baseline to 6 months | 6 months
  The OHS is a 12-item patient-reported outcome measure designed to assess hip function and pain within the last four weeks among patients suffering from hip osteoarthritis in one score. The total score ranges from 0 to 48, with higher scores indicating better disease status.

SECONDARY OUTCOMES:
Change in the Hip disability and Osteoarthritis Outcome Score (HOOS) pain subscale from baseline to 6 months | 6 months
  The HOOS pain subscale is a 10-item patient-reported outcome measure designed to assess hip pain in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better pain status.
Change in the HOOS symptoms subscale from baseline to 6 months | 6 months
  The HOOS pain subscale is a five-item patient-reported outcome measure designed to assess other hip symptoms in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better symptoms status.
Change in the HOOS activities of daily living (ADL) function subscale from baseline to 6 months | 6 months
  The HOOS ADL function subscale is a 17-item patient-reported outcome measure designed to assess ADL function in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better ADL function status.
Change in the HOOS quality-of-life subscale from baseline to 6 months | 6 months
  The HOOS quality-of-life subscale is a four-item patient-reported outcome measure designed to assess hip-related quality-of-life in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better quality-of-life status.
Change in the HOOS sports and recreation subscale from baseline to 6 months | 6 months.
  The HOOS sports and recreation subscale is a four-item patient-reported outcome measure designed to assess sports and recreation function in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better sports and recreation status.
Change in the University of California Los Angeles (UCLA) Activity Score | 6 months
  The UCLA Activity Score is a single-item patient-reported outcome measure designed to assess physical activity level. The score ranges from 1 to 10, with higher scores indicating greater physical activity level.
Change in the 40 metre Fast Paced Walk Test (40m-FPWT) from baseline to 6 months | 6 months
  The 40m-FPWT is a physical function test designed to assess short distance maximum walking speed (meters/second).
Change in the 30 second Chair Stand Test (30s-CST) from baseline to 6 months | 6 months
  The 30s-CST is a physical function test designed to assess sit-to-stand function (number of repetitions).
Number of Serious Adverse Events (SAE) from baseline to 6 months | 6 months.
  SAE according to the International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) guidelines will be collected from The Danish National Patient Registry and medical record review conducted at the 6 months follow-up. Furthermore, a short patient-reported questionnaire at the 3 and 6 months follow-up will be used to ensure that all SAE are recorded.

OTHER OUTCOMES:
Change in hip pain intensity on a 101-point Visual Analogue Scale (VAS) from baseline to 6 months | 6 months
  The VAS pain is a single-item patient-reported outcome measure used to assess mean hip pain intensity at rest, and main hip pain intensity activity during the previous 24 hours. The total scale ranges from 0 (no pain) to 100 (worst pain imaginable).
Change in EuroQol Group 5-dimension 5-level (EQ-5D-5L) from baseline to 6 months | 6 months
  The EQ-5D-5L is a five-item patient-reported outcome measure designed to assess generic health-related quality-of-life. The total score of the descriptive index and EQ-VAS ranges from -0.624 (worst) to 1.000 (best) and 0 (worst imaginable health) to 100 (best imaginable health), respectively. This will also allow for a later cost-utility analysis.
Change in number of patients using pain medication related to the hip from baseline to 6 months | 6 months
  Medicine consumption will be assessed with the following question: "Have you been taking pain medication within the last week?" on a dichotomous scale (yes/no). Patients answering "yes" will be asked to provide type of medication on a categorical scale (Paracetamol, NSAID, morphine/opioids, Gabapentin, and other), frequency on 6-point Likert-scale ranging from "1 time a week" to "4 times a day or above", and asked "Have you primarily been taking pain medication due to your hip?" rated on a dichotomous scale (yes/no). Patients responding "no" to the latter question will be asked "If no, have you been taking pain medication due to other known diseases or disorders?" rated on on a dichotomous scale (yes/no).
Global Perceived Effect (GPE) at 6 months | 6 months
  The GPE of the interventions will be assessed for seven domains, including overall hip problems, hip pain, hip symptoms, ADL function, sports and recreation, hip-related quality-of-life, and physical activity on a 15-point Likert scale ranging from "a very great deal worse" (worst) to "a very great deal better" (best).
Patient Acceptable Symptom State (PASS) at 6 months | 6 months
  PASS will be assessed with the following question: "When you think of your hip function, will you consider your current condition as satisfying?" By hip function, you should take into account your activities of daily living, sport and recreational activities, your hip pain and other symptoms and your quality-of-life on a dichotomous scale (yes/no).
Treatment Failure at 6 months | 6 months
  Patient-reported treatment failure will be assessed only by patients answering "no" to PASS with the following question: "Would you consider your current state as being so unsatisfactory that you think the treatment has failed?" on a dichotomous scale (yes/no).
Change in physical activity (tri-axial accelerometer) from baseline to 6 months | 6 months
  Physical activity will be recorded with a tri-axial accelerometer (AX3, Axivity, Ltd., Newcastle, UK) mounted on the lateral thigh during a 7 day period. Data will be post-processed using a custom designed algorithm (MATLAB, Mathworks, Natick, MA, USA).
Change in isometric hip muscle strength from baseline to 6 months | 6 months
  Isometric muscle strength of the index hip will be recorded for hip extension, flexion, and abduction with a handheld dynamometer (Commander Echo Wireless Console and Muscle Tester, JTECH Medical, Salt Lake City, Utah, USA) and reported as Newton meters per kilogram of the bodyweight (Nm/kg).
Number of total hip arthroplasty surgeries from baseline to 6 months (PRT group) | 6 months
  Number of total hip arthroplasty surgeries performed in the PRT group will be registered through a medical record review.
Number of PRT sessions from baseline to 3 months (PRT group) | 3 months
  In the PRT group, the number of PRT sessions participated in by the patient will be registered by the supervising physiotherapist. High compliance will be defined as participation in ≥75% of the training sessions corresponding to 18 out of 24 sessions; moderate compliance as participation in 50-74% of the sessions; and poor compliance as participation in <50% of the sessions.
Change in training load from baseline to 3 months (PRT group) | 3 months
  Training load of each exercise in the PRT group will be registered by the supervising physiotherapist and reported as kilogram (kg).
Number of patients performing unsupervised exercise from 3 to 6 months (PRT group) | 3 months
  Following the 12-week supervised PRT program, adherence to three-months of optional unsupervised PRT will be measured by a patient-reported questionnaire.
Number of patients receiving supervised postoperative rehabilitation from baseline to 6 months (THA group) | 6 months
  Participation in postoperative supervised exercise in the THA group will be assessed using a patient-reported questionnaire.
Number of patients receiving other treatments from baseline to 6 months. | 6 months
  Other treatments related to the index hip will be assessed using a patient-reported questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frydendal, PT, MSc, Principal Investigator — Vejle Hospital and University of Southern Denmark; Søren Overgaard, Prof., MD, Study Director — Odense University Hospital and University of Southern Denmark; Inger Mechlenburg, Prof., DMSc, Study Chair — Aarhus University Hospital and Aarhus University; Kim Gordon Ingwersen, PT, PhD, Study Chair — Vejle Hospital and University of Southern Denmark; Lone Ramer Mikkelsen, PT, PhD, Study Chair — Silkeborg Regional Hospital; Robin Christensen, Prof., PhD, Study Chair — The Parker Institute and Odense University Hospital; Claus Varnum, PhD, MD, Study Chair — Vejle Hospital; Henrik Morville Schrøder, PhD, MD, Study Chair — Naestved Hospital
Locations (4):
- Denmark (4):
  - Department of Orthopaedic Surgery, Aarhus University Hospital (AUH), Aarhus
  - Department of Orthopaedic Surgery, Naestved Hospital, Næstved
  - Department of Orthopaedic Surgery and Traumatology, Odense University Hospital (OUH), Odense
  - Depatment of Orthopaedic Surgery, Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: Yes
Anonymised patient-level data for the primary and all secondary outcome measures will be made available if required by the scientific journal, in which the results of the trial are published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after publication of the trial.
Access Criteria: Data access will be reviewed by the author group. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Bryld ES, Christiansen L, Ingwersen KG, Overgaard S, Mikkelsen LR, Mechlenburg I, Frydendal T. Training load and pain response during progressive resistance training in patients with hip osteoarthritis in the PROHIP trial. Osteoarthr Cartil Open. 2025 Oct 4;7(4):100690. doi: 10.1016/j.ocarto.2025.100690. eCollection 2025 Dec. PMID 41141645
- [Derived] Frydendal T, Christensen R, Mechlenburg I, Mikkelsen LR, Varnum C, Graversen AE, Kjaersgaard-Andersen P, Revald PH, Hofbauer C, Bieder MJ, Qassim H, Munir MS, Jakobsen SS, Nielsen SM, Ingwersen KG, Overgaard S. Total Hip Replacement or Resistance Training for Severe Hip Osteoarthritis. N Engl J Med. 2024 Oct 31;391(17):1610-1620. doi: 10.1056/NEJMoa2400141. PMID 39476341
- [Derived] Frydendal T, Thomsen KS, Mechlenburg I, Mikkelsen LR, Overgaard S, Ingwersen KG, Myburgh C. Patient and public involvement to inform the protocol of a clinical trial comparing total hip arthroplasty with exercise: an exploratory qualitative case study. BMJ Open. 2023 Apr 24;13(4):e070866. doi: 10.1136/bmjopen-2022-070866. PMID 37094895
- [Derived] Frydendal T, Christensen R, Mechlenburg I, Mikkelsen LR, Overgaard S, Ingwersen KG. Total hip arthroplasty versus progressive resistance training in patients with severe hip osteoarthritis: protocol for a multicentre, parallel-group, randomised controlled superiority trial. BMJ Open. 2021 Oct 22;11(10):e051392. doi: 10.1136/bmjopen-2021-051392. PMID 34686555

DOCUMENTS (3):
  • Statistical Analysis Plan: Statistical Analysis Plan: RCT (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT04070027/SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan: Generalizability (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT04070027/SAP_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan: Physical Activity (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT04070027/SAP_003.pdf